CLINICAL TRIAL: NCT03257241
Title: A PALG Prospective Multicenter Clinical Trial to Compare the Efficacy of Two Standard Induction Therapies (DA-90 vs DAC) and Two Standard Salvage Regimens (FLAG-IDA vs CLAG-M) in AML Patients ≤ 60 Years Old
Acronym: PALG-AML1/2016
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polish Adult Leukemia Group (Other)
Responsible Party: Principal Investigator, Agnieszka Wierzbowska, Study Coordinator, Polish Adult Leukemia Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALG-AML1/2016
Record Dates: First submitted 2017-08-04; First posted 2017-08-22 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: aml; acute myeloid leukemia; DAC; DA-90; FLAG-IDA; CLAG-M; Ara-C; HiDAC
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Daunorubicin; Cytarabine; Decitabine; Cladribine; Mitoxantrone; Granulocyte Colony-Stimulating Factor; fludarabine; Idarubicin

STUDY DESIGN:
Intervention Model Description: Comparison of the efficacy of two standard induction treatment protocols (DA-90 and DAC) in patients with newly-diagnosed AML (with the exception of acute promyelocytic leukemia). Comparison of the efficacy of two standard reinduction treatment protocols (CLAG-M and FLAG-IDA) in patients with refractory and relapsed AML.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A arm (DA-90) (Active Comparator): Induction I:
  * DNR 90 mg/m2 D 1-3 in 30-60 min i.v. infusion
  * Ara-C 100 mg/m2 D 1-7 in 24 h i.v. infusion
  Interventions: Drug: A arm (DA-90)
- B arm (DAC) (Active Comparator): Induction I:
  * DNR 60 mg/m2 D 1-3 in 30-60 min i.v. infusion
  * cladribine 5 mg/m2 D 1-5 in 2 h i.v. infusion prior to Ara-C
  * Ara-C 200 mg/m2 D 1-7 in 22 h i.v. infusion.
  Interventions: Drug: B arm (DAC)
- A arm (CLAG-M) (Active Comparator): Cladribine 5mg/m2 in 2 h i.v. infusion on days (1-5) Ara-C 2 g/m2 in 4 h i.v. infusion, 2 h after cladribine infusion on days (1-5) Mitoxantrone 10 mg/m2 i.v. 1xd on days (1-3) G-CSF 30MU s.c. 1xd from day 0 to 5 of the treatment (6 doses).
  Interventions: Drug: A arm (CLAG-M)
- B arm (FLAG-IDA) (Active Comparator): Fludarabine 30 mg/m2 in 30-min i.v. infusion on days (1-5) Ara-C 2 g/m2 in 4 h i.v. infusion, 2 h after fludarabine infusion on days (1-5). Idarubicin 8 mg/m2 i.v. 1xd on days (1-3) G-CSF 30MU s.c. 1xd from day 0 to 5 of the treatment (6 doses).
  Interventions: Drug: B arm (FLAG-IDA)

INTERVENTIONS:
Drug: A arm (DA-90) — After confirming the diagnosis, assuming the inclusion criteria and exclusion criteria are respected, the patients are randomized to one of two standard induction treatment protocols (A arm: DA-90 vs B arm: DAC). After completing induction I, an early bone marrow assessment is performed on day 14 from the beginning of the treatment (+ day 7 after finishing chemotherapy) using the cytological method and MRD is assessed by the immunophenotyping method. Therapeutic decision is taken on the basis of the cytological assessment. Patients, in whom the percentage of blasts in the bone marrow on day 14 is > 10%, receive early induction II from day 16. An Immunophenotype test is a complementary examination.
  Other Names: Daunorubicin, Cytarabine
  Arms: A arm (DA-90)
Drug: B arm (DAC) — After confirming the diagnosis, assuming the inclusion criteria and exclusion criteria are respected, the patients are randomized to one of two standard induction treatment protocols (A arm: DA-90 vs B arm: DAC). After completing induction I, an early bone marrow assessment is performed on day 14 from the beginning of the treatment (+ day 7 after finishing chemotherapy) using the cytological method and MRD is assessed by the immunophenotyping method. Therapeutic decision is taken on the basis of the cytological assessment. Patients, in whom the percentage of blasts in the bone marrow on day 14 is > 10%, receive early induction II from day 16. An Immunophenotype test is a complementary examination.
  Other Names: Daunorubicin, Cladribine, Cytarabine
  Arms: B arm (DAC)
Drug: A arm (CLAG-M) — Patients who do not achieve CR after two courses of induction therapy or patients with relapsed leukemia are eligible for emergency treatment ("salvage") according to the CLAG- M or FLAG-IDA protocol.
  Other Names: Cladribine, Cytarabine, Mitoxantrone, G-CSF
  Arms: A arm (CLAG-M)
Drug: B arm (FLAG-IDA) — Patients who do not achieve CR after two courses of induction therapy or patients with relapsed leukemia are eligible for emergency treatment ("salvage") according to the CLAG- M or FLAG-IDA protocol.
  Other Names: Fludarabine, Cytarabine, Idarubicin, G-CSF
  Arms: B arm (FLAG-IDA)

SUMMARY:
The study will include newly-diagnosed AML patients, not suffering acute promyelocytic leukemia; aged 18-60 years, who are eligible for standard induction chemotherapy. The patients will be randomized to one standard induction regimen (DAC or DA-90). At day seven after completion of induction, a bone marrow aspiration with MRD will be performed for an early evaluation of response to treatment. Patients without bone marrow blast reduction below 10% at day seven after induction will be given a second early induction course. Patients who do not achieve CR after two induction courses will be randomized to one of the standard salvage regimens (FLAG-IDA or CLAG-M). Postremission treatment intensity will be adjusted to risk group based on cytogenetic and molecular risk factors at diagnosis and AML biology (secondary AML, therapy related AML). Patients with a low risk of relapse will be allocated to consolidation, with three courses of high doses of Ara-C (HiDAC), or two courses of HiDAC with subsequent autologous stem cell transplantation. Intermediate- or high-risk patients will be referred for allogeneic stem cell transplantation, if they have a matched donor. Until transplantation, consolidation with HiDAC will be continued.

DETAILED DESCRIPTION:
The successful treatment of acute myeloid leukemia (AML) depends on the ability to achieve complete remission (CR) and to prevent relapse. Both may be affected by the efficacy of induction chemotherapy. The gold standard for treatment since 1982 has been DA, a regimen of three days of daunorubicin (DNR) and seven days of cytarabine (Ara-C) which results in complete remission in 50 to 75% of patients; this is typically administered intravenously, with daunorubicin administered at a dose of 45 mg per square meter of body-surface area daily for three days, and cytarabine given at a dose of 100 mg per square meter daily for seven days. Neither substituting DNR with another anthracycline nor the addition of thioguanine or etoposide has been demonstrated to improve outcome. Recently it has been proved that high-dose daunorubicin (90 mg/m2) in induction (DA-90) resulted in a higher rate of complete remission (70.6% vs. 57.3%, P<0.001) and improved overall survival (median, 23.7 vs. 15.7 months; P = 0.003) without any increase in serious adverse events, compared with the standard dose of the drug.

An alternative method to intensify induction treatment is by the addition of the purine analog cladribine. Cladribine was demonstrated to increase cellular uptake of Ara-C and accumulation of Ara-CTP in leukemic blasts by 50% to 65% and to have direct antileukemic activity based on incorporation of metabolites into the DNA of proliferating cells. In two randomized trials by the Polish Adult Leukemia Group (PALG), the investigators demonstrated that the combination of cladribine with DNR (60 mg/m2) and Ara-C (DAC) resulted in a significantly increased CR rate after a single induction course compared with the standard two-drug induction (DA-60). The DAC arm was found to have a survival advantage over the DA-60 arm for patients aged 50 years or older (P =. 005), those with an initial leukocyte count above 50G /L (P < .03), and those with an unfavorable karyotype (P < .03). Both induction protocols have the same level of recommendation by the National Cancer Comprehensive Network (NCCN) for routine use (level I), and are commonly used for the treatment of newly diagnosed AML in Poland.

As no randomized comparison of these two standard protocols has yet been performed, the aim of the proposed study is to compare the efficacy of these two standard induction protocols in terms of achievement of CR, early leukemia elimination (at day seven, post induction) and quality of remission measured by minimal residual disease level. Additionally, overall survival (OS), event-free survival (EFS) and disease-free survival (DFS) will be analyzed. It is also intended to compare the hematological and non-hematological toxicity of both regimens.

However, in younger adults with AML treated with standard induction chemotherapy, 20-35% do not achieve CR and 50-70% with CR may be expected to relapse within three years. Patients with primary refractory disease and with relapses following CR1 have a significantly poorer outcome. The optimum strategy at the time of relapse or for patients with refractory disease remains uncertain. Allogeneic transplantation can be curative for the minority of patients who achieve second CR (2CR) and for whom a suitable donor is available. For the majority of patients, additional chemotherapy is given in the hope of achieving remission. Most salvage therapies utilize high or intermediate doses of arabinoside cytosine (Ara-C) in combination with other agents to overcome resistance in leukemic cells. Previous studies have shown that a combination of the purine analog fludarabine (FA) and cytosine arabinoside (Ara-C) increases the accumulation of Ara-C-5' triphosphate (Ara-CTP) responsible for the cytotoxic effect in leukemic blasts. This combination of FA plus Ara-C was initially explored in refractory and relapsed AML patients with satisfactory results. It is also likely that these results can be improved by the addition of granulocyte-colony stimulating factor (G-CSF). Such a combination of FA, Ara-C, idarubicin and G-CSF (the FLAG-IDA regimen) has been used in the treatment of refractory and relapsed AML and poor prognosis myelodysplastic syndromes (MDS), with CR rates of between 30-80% being reported. Recent studies have shown that another purine analog, cladribine (2-CdA), is also able to enhance Ara-CTP accumulation in leukemic blasts and that the combination of 2-Cda with Ara-C exhibited synergistic effect on inhibition of myeloid leukemic cell proliferation, induction of apoptosis, and on disruption of mitochondrial membrane potential.

Two previous PALG studies have confirmed that the CLAG-M regimen (a combination of cladribine, Ara-C, G-CSF and mitoxantrone) has high efficacy and low toxicity in refractory/relapsed AML patients. This salvage regimen was particularly effective in a very poor-risk subgroup with primary refractoriness, early relapse or relapse after stem cell transplantation. Both salvage protocols, CLAG-M and FLAG-Ida, are wildly used in the treatment of relapsed/refractory AML and both have the highest level of NCCN recommendation. However, these two standard salvage protocols have yet to be examined as part of any randomized study. Therefore, the aim of this study is to compare the efficacy of these two standard reinduction protocols (CLAG-M vs FLAG-IDA) in terms of achievement of CR, and quality of remission measured by minimal residual disease level. Additionally, the overall survival (OS), event-free survival (EFS) and disease-free survival (DFS) will be analyzed. The study will also compare the hematological and non-hematological toxicity of both regimens.

The study will include newly-diagnosed AML patients, not suffering acute promyelocytic leukemia; aged 18-60 years, who are eligible for standard induction chemotherapy. The patients will be randomized to one standard induction regimen (DAC or DA-90). At day seven after completion of induction, a bone marrow aspiration with MRD will be performed for an early evaluation of response to treatment. Patients without bone marrow blast reduction below 10% at day seven after induction will be given a second early induction course. Patients who do not achieve CR after two induction courses will be randomized to one of the standard salvage regimens (FLAG-IDA or CLAG-M). Postremission treatment intensity will be adjusted to risk group based on cytogenetic and molecular risk factors at diagnosis and AML biology (secondary AML, therapy related AML). Patients with a low risk of relapse will be allocated to consolidation, with three courses of high doses of Ara-C (HiDAC), or two courses of HiDAC with subsequent autologous stem cell transplantation. Intermediate- or high-risk patients will be referred for allogeneic stem cell transplantation, if they have a matched donor. Until transplantation, consolidation with HiDAC will be continued.

The primary end point of the study is CR rate after one and two induction courses. The secondary end-points are the quality of CR (MRD), OS, DFS, PFS, CR rate after salvage regimen.

It is planned to include 582 patients with newly-diagnosed AML. This will allow a 10% difference in CR rate between DAC and DA-90 induction regimens to be confirmed with a power of 80% and level of significance 0.05.

The study includes neither any experimental drug nor procedures that are not of the standard of treatment for AML.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute myeloid leukemia (≥20% of blasts in the bone marrow)
2. Previously untreated AML

   * AML de novo
   * AML secondary to the myelodysplastic syndromes (MDS)
   * AML secondary towards used therapies or agents, which can induce leukemia (e.g., irradiation, alkylating drugs, topoisomerase II inhibitors) with a primary tumor in remission for at least 2 years.
3. Age ≥ 18 years and ≤60 years while signing a written consent form
4. A clinical condition allowing induction treatment to be performed

   * General state according to the ECOG ≤ 2 scale (Annex 1)
   * Index of comorbidities, HCT-CI ≤ 3, according to Sorror et al. (43) (Annex 2)
5. Normal function of the liver and kidneys defined as:

   * Bilirubin of ≤1.5 of the upper limit of the normal range
   * ALT ≤2.5 x of the upper limit of the normal range
   * AST ≤2.5 x of the upper limit of the normal range
   * Creatinine ≤1.5 of the upper limit of the normal range
6. A negative pregnancy test result in women of reproductive age, or women after menopause
7. The patient has understood and signed an informed consent form (Annex 3)
8. The patient has given consent to adhere to scheduled appointments in the study and the remaining protocol requirements.

Exclusion Criteria:

1. Diagnosis or suspicion of acute promyelocytic leukemia (APL)
2. Lack of consent for participation in the study
3. Active cancerous disease other than AML (with the exception of carcinoma basocellulare cutis)
4. Diagnosis of unstable angina pectoris, significant cardiac arrhythmia or class III or IV congestive heart failure according to the New York Heart Association (NYHA) functional classification
5. Pregnancy
6. Uncontrolled mycotic, bacterial or viral systemic infection
7. Active HIV, or hepatitis B or C virus infection
8. The use of another form of experimental therapy within 28 days of the commencement of treatment
9. The presence of another comorbidity or improper study results which could expose the patient to excessive hazard (HCT-CI>3)
10. Any other serious health disorders, abnormal results of laboratory tests or mental disorders which would interfere with participation in the study
11. The presence of other comorbidities which would disturb the interpretation of the data obtained in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 582 (Estimated)
Dates: Start 2017-07-03 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Induction regimen efficacy (DA-90 vs DAC) - I induction | On +7 day after chemotherpay
  Comparison of total remission rates after 1 induction course of DA-90 and DAC.
Induction regimen efficacy (DA-90 vs DAC) - II induction | On +28 day after chemotherapy or after complete morphology regeneration (if it occurs before day +28)
  Comparison of total remission rates after II induction course of DA-90 and DAC.
Salvage regimen efficacy (CLAG-M vs FLAG-IDA) - I reinduction | On +28 day after chemotherapy or after complete morphology regeneration (if it occurs before day +28)
  Comparison of total remission rates after I reinduction course of CLAG-M and FLAG-IDA
Salvage regimen efficacy (CLAG-M vs FLAG-IDA) - II reinduction | On +28 day after chemotherapy or after complete morphology regeneration (if it occurs before day +28)
  Comparison of total remission rates after II reinduction course of CLAG-M and FLAG-IDA

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Giebel, Prof., Principal Investigator — Polish Adult Leukemia Group
Locations (10):
- Weill Cornell Medicine, New York, New York, United States
- Poland (9):
  - Medical University of Bialystok Clinical Hospital, Bialystok
  - Markiewicz Memorial Oncology Center Brzozow, Brzozów
  - University Clinical Centre in Gdansk, Gdansk
  - Holycross Cancer Center, Kielce
  - Ludwik Rydygier Memorial Specialized Hospital, Krakow
  - Regional Specialised Hospital in Legnica, Legnica
  - Copernicus Memorial Hospital in Lodz Comprehensive Cancer Center and Traumatology, Lodz
  - Independent Public University Hospital No. 1 in Lublin, Lublin
  - Clinical Hospital at the Karol Marcinkowski Medical University in Poznan, Poznan